CLINICAL TRIAL: NCT03634943
Title: Evaluation of Nutritional Practices in the Critical Care Patient at the Intensive Care Unit
Brief Title: Evaluation of Nutritional Practices in the Critical Care
Acronym: ENPIC
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Arnau de Vilanova (Other); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Juan Carlos Lopez-Delgado, PhD, Intensive Care Specialist, Hospital Universitari de Bellvitge
Other Study IDs: PR401/17
Record Dates: First submitted 2018-08-12; First posted 2018-08-17 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Nutritional Support; Intensive Care Unit; Critical Illness
Keywords: Clinical Practice Guidelines
MeSH Terms: conditions — Critical Illness | interventions — Nutritional Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Nutritional Support: Patients expected to be admitted >72h at the Intensive Care Unit with the need of artificial Nutritional Support
  Interventions: Other: Patients with Nutritional Support

INTERVENTIONS:
Other: Patients with Nutritional Support — Evaluation of Enteral Nutrition or Parenteral Nutrition or both administered to the patients needing artificial Nutritional Support

SUMMARY:
Background: The adequacy of the artificial Nutritional Support (NS) in the critical care patient has implications in morbidity and prognosis. Clinical practice guidelines (CPG) are an important tool for healthcare professionals in their daily practice and a method of consultation for the correct treatment of patients. Also, the evidence remains low and there are important controversies regarding the NS in the critical care patient.

Hypothesis: The NS generates great controversy in the professionals involved in the care of critical care patients due to the contradictory results in literature. Despite this, the CPG should serve to standardize the treatment of patients and provide a better adherence to current knowledge in this setting. The importance of NS is underestimated and there is a need to perform proper evaluation of the impact of nutrition.

Objectives: To evaluate and analyze NS practices in critically ill patients in different ICUs and assess the adherence to CPGs. To evaluate the relationship of nutrition and outcomes in the ICU.

Methodology: Prospective multicenter observational study. Collection of variables from different participating ICUs and the characteristics of the NS of the different admitted patients. Monitoring of nutritional practices and complications. Evaluation of outcomes (e.g. mortality, ICU complications, etc.) with NS.

Expected results: Better understanding of the NS and its impact on morbidity and mortality; development of strategies to reduce low adherence to CPGs, improving the quality of care associated with this field in critical care patients; obtain clinical information that will serve as a basis for conducting intervention studies.

DETAILED DESCRIPTION:
Methods (additional information): The NS (Nutritional Support) in the ICUs will be administered according to the usual practice of the medical and nursing staff and to the protocols established in each unit. The rate of initiation, the dose of macronutrients and the increase in contributions will be made according to the criteria of each participating ICU and the responsible physician (including the use of prokinetics or parenteral nutrition).

All the complications described associated with the artificial Nutritional support and others related to the critical patient will be evaluated daily by the research team and reflected in the electronic data collection form (eCRF).

The eCRF has been carried out through the REDCAP ™ platform and designed by the Department of Information Technology of Lleida of the Universitari Arnau de Vilanova Hospital, under the supervision of Dr. Lluís Servià, principal investigator of the present project. The responsible of the computer centre is Joan Escobar-Ortiz. The data will be stored in a server of the center and will be coded to comply with the confidentiality of the same and for a correct anonymization of patients based on Regulatory Laws.

The study has the approval of each ethics committee of each participating centre.

Statistical analyses will be performed by the department of statistics of University of Lleida under close supervision of Javier Trujillano-Cabello and the principal investigators of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Need of ICU admission >72h.
* Need of Artificial Nutrional Support (Enteral Nutrition or Parenteral Nutrition or both).

Exclusion Criteria:

* Not specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Critical Care patients needing Artificial Nutritional Support
Sampling Method: Non-Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Kilocalories delivered by enteral and/or parenteral route and Energy balance | Daily to a maximum of 14 days after Intensive Care Unit Admission
  Kilocalories delivered by nutritional support - (minus) nutritional support target in Kilocalories
gram of proteins delivered by enteral and/or parenteral route | Daily to a maximum of 14 days after Intensive Care Unit Admission
  Proteins delivered by nutritional support - (minus) nutritional support target in gram of proteins
Rate of complications related with nutritional support (Enteral and/or Parenteral route) | Daily to a maximum of 14 days after Intensive Care Unit Admission
  Main artificial nutritional support serious complications (i.e. constipation, higher residual gastric volume, vomiting, diarrhea associated with enteral nutrition, meseteric ischemia) requiring a therapeutical intervention or modification of the nutritional support - safety related variable
Rate of 28-day mortality associated with the characteristics of nutritional support (e.g., gram of proteins, etc.) | Daily to a maximum of 28 days after Intensive Care Unit Admission
  Influence of nutritional support or any nutrition-related variable on mortality during ICU admission

SECONDARY OUTCOMES:
Time from Intensive Care Unit admission to the start of enteral nutrition | Up to 120 hours after Intensive Care Unit Admission
  Time frame in hours from Intensive Care Unit admission to the start of enteral nutrition
Dose of vasoactive drugs | Daily to a maximum of 14 days after Intensive Care Unit Admission
  Dose of vasoactive drugs (highest daily), in μg/kg/min
Glycaemic control | Daily to a maximum of 14 days after Intensive Care Unit Admission
  Daily measurement of maximum and minimum glucose

CONTACTS AND LOCATIONS:
Overall Officials: Teodoro Grau-Carmona, Ph.D., Principal Investigator — Hospital 12 de Octubre; Lluís Servia-Goixart, Ph.D., Principal Investigator — Hospital Arnau de Vilanova / Biomedical Research Institute of Lleida (IRBLleida) Institut de Recerca Biomèdica de Lleida; Juan Carlos Lopez-Delgado, Ph.D, Principal Investigator — Hospital Universitari de Bellvitge
Locations (43):
- Spain (43):
  - Hospital Sant Joan d' Alacant, Sant Joan d'Alacant, Alicante
  - H. Manacor, Manacor, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - H. General de Granollers, Granollers, Barcelona
  - Hospital Universitari de Bellvitge (Cardiology Unit), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Mutua Terrasa., Terrassa, Barcelona
  - Hospital General Universitario de Castellón, Castellon, Castellón
  - Hospital Universitario de Puerto Real, Puerto Real, Cádiz
  - Hospital de Barbastro, Barbastro, Huesca
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Quirón Sur, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Infanta Cristina, Parla, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Plató, Barcelona
  - Hospital de la Santa Creu i Sant Pau., Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitari Josep Trueta, Girona
  - Hospital General San Jorge, Huesca
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario 12 de Octubre (Trauma Unit), Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital General Universitario Reina Sofia, Murcia
  - Hosptial General Universitario Morales Meseguer, Murcia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari Doctor Peset, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Rio Hortega, Valladolid
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
  - Hospital Royo Villanova, Zaragoza

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed by the principal investigators of each participating hospital. Share IPD is not allowed in the present study to other researchers.

REFERENCES:
- [Result] Marik PE, Zaloga GP. Early enteral nutrition in acutely ill patients: a systematic review. Crit Care Med. 2001 Dec;29(12):2264-70. doi: 10.1097/00003246-200112000-00005. PMID 11801821
- [Result] Heyland D, Cook DJ, Winder B, Brylowski L, Van deMark H, Guyatt G. Enteral nutrition in the critically ill patient: a prospective survey. Crit Care Med. 1995 Jun;23(6):1055-60. doi: 10.1097/00003246-199506000-00010. PMID 7774216
- [Result] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Result] Dvir D, Cohen J, Singer P. Computerized energy balance and complications in critically ill patients: an observational study. Clin Nutr. 2006 Feb;25(1):37-44. doi: 10.1016/j.clnu.2005.10.010. PMID 16321459
- [Result] Deitch EA. Role of the gut lymphatic system in multiple organ failure. Curr Opin Crit Care. 2001 Apr;7(2):92-8. doi: 10.1097/00075198-200104000-00007. PMID 11373517
- [Result] Harvey SE, Parrott F, Harrison DA, Bear DE, Segaran E, Beale R, Bellingan G, Leonard R, Mythen MG, Rowan KM; CALORIES Trial Investigators. Trial of the route of early nutritional support in critically ill adults. N Engl J Med. 2014 Oct 30;371(18):1673-84. doi: 10.1056/NEJMoa1409860. Epub 2014 Oct 1. PMID 25271389
- [Result] Patel JJ, Codner P. Controversies in Critical Care Nutrition Support. Crit Care Clin. 2016 Apr;32(2):173-89. doi: 10.1016/j.ccc.2015.11.002. Epub 2016 Feb 4. PMID 27016160
- [Result] Artinian V, Krayem H, DiGiovine B. Effects of early enteral feeding on the outcome of critically ill mechanically ventilated medical patients. Chest. 2006 Apr;129(4):960-7. doi: 10.1378/chest.129.4.960. PMID 16608945
- [Result] Flordelis Lasierra JL, Perez-Vela JL, Montejo Gonzalez JC. Enteral nutrition in the hemodynamically unstable critically ill patient. Med Intensiva. 2015 Jan-Feb;39(1):40-8. doi: 10.1016/j.medin.2014.04.002. Epub 2014 Jun 4. English, Spanish. PMID 24907000
- [Result] Arabi YM, Aldawood AS, Haddad SH, Al-Dorzi HM, Tamim HM, Jones G, Mehta S, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Afesh L; PermiT Trial Group. Permissive Underfeeding or Standard Enteral Feeding in Critically Ill Adults. N Engl J Med. 2015 Jun 18;372(25):2398-408. doi: 10.1056/NEJMoa1502826. Epub 2015 May 20. Erratum In: N Engl J Med. 2015 Sep 24;373(13):1281. doi: 10.1056/NEJMx150028. PMID 25992505
- [Result] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Result] Wischmeyer PE. Are we creating survivors...or victims in critical care? Delivering targeted nutrition to improve outcomes. Curr Opin Crit Care. 2016 Aug;22(4):279-84. doi: 10.1097/MCC.0000000000000332. No abstract available. PMID 27327244
- [Result] Wei X, Day AG, Ouellette-Kuntz H, Heyland DK. The Association Between Nutritional Adequacy and Long-Term Outcomes in Critically Ill Patients Requiring Prolonged Mechanical Ventilation: A Multicenter Cohort Study. Crit Care Med. 2015 Aug;43(8):1569-79. doi: 10.1097/CCM.0000000000001000. PMID 25855901
- [Derived] Lopez-Delgado JC, Servia-Goixart L, Grau-Carmona T, Bordeje-Laguna L, Portugal-Rodriguez E, Lorencio-Cardenas C, Vera-Artazcoz P, Macaya-Redin L, Martinez-Carmona JF, Marin Corral J, Flordelis-Lasierra JL, Seron-Arbeloa C, Alcazar-Espin MLN, Navas-Moya E, Aldunate-Calvo S, Nieto Martino B, Martinez de Lagran I. Factors associated with the need of parenteral nutrition in critically ill patients after the initiation of enteral nutrition therapy. Front Nutr. 2023 Aug 24;10:1250305. doi: 10.3389/fnut.2023.1250305. eCollection 2023. PMID 37693244
- [Derived] Servia-Goixart L, Lopez-Delgado JC, Grau-Carmona T, Trujillano-Cabello J, Bordeje-Laguna ML, Mor-Marco E, Portugal-Rodriguez E, Lorencio-Cardenas C, Montejo-Gonzalez JC, Vera-Artazcoz P, Macaya-Redin L, Martinez-Carmona JF, Iglesias-Rodriguez R, Monge-Donaire D, Flordelis-Lasierra JL, Llorente-Ruiz B, Menor-Fernandez EM, Martinez de Lagran I, Yebenes-Reyes JC; ENPIC Study Investigators. Evaluation of Nutritional Practices in the Critical Care patient (The ENPIC study): Does nutrition really affect ICU mortality? Clin Nutr ESPEN. 2022 Feb;47:325-332. doi: 10.1016/j.clnesp.2021.11.018. Epub 2021 Nov 16. PMID 35063222